CLINICAL TRIAL: NCT03846505
Title: Oxytocin to Enhance Alcohol Behavioral Couple Therapy (ABCT)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Julianne Flanagan, Associate Professor, Department of Psychiatry and Behavioral Sciences, Addiction Sciences, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00082233; 1R01AA027212 (NIH)
Record Dates: First submitted 2019-02-17; First posted 2019-02-19 (Actual); Results first posted 2025-02-21 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-01

CONDITIONS: Alcohol Use Disorder; Couples
Keywords: Couple; Alcohol; Therapy
MeSH Terms: conditions — Alcoholism | interventions — Oxytocin; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Oxytocin and Therapy Placebo and Therapy
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Oxytocin (Experimental): A 40-IU dose of oxytocin will be self-administered 30 minutes prior to the start of each weekly ABCT session.
  All participants will receive 12 weekly, 90-minute ABCT therapy sessions delivered by trained Masters or Doctoral-level clinicians consistent with the published manual.
  Interventions: Drug: Oxytocin
- Placebo (Placebo Comparator): A placebo will be self-administered 30 minutes prior to the start of each weekly ABCT session.
  All participants will receive 12 weekly, 90-minute ABCT therapy sessions delivered by trained Masters or Doctoral-level clinicians consistent with the published manual.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Oxytocin — A 40-IU dose of oxytocin will be self-administered 30 minutes prior to the start of each weekly ABCT session.
  Other Names: Pitocin
  Arms: Oxytocin
Other: Placebo — A placebo will be self-administered 30 minutes prior to the start of each weekly ABCT session.
  Other Names: Saline
  Arms: Placebo

SUMMARY:
Alcohol Behavioral Couples Therapy (ABCT) is a manualized 12-session, weekly psychosocial intervention that simultaneously reduces alcohol use disorder (AUD) severity and improves relationship functioning. However, there remains room to improve ABCT outcomes. A growing literature suggests that intranasal oxytocin is a medication that holds promise to achieve that goal. Oxytocin has demonstrated the ability to increase prosocial behavior (e.g., trust, safety, social cognition) and restore sensitivity to natural rewards such as interpersonal relationships that are commonly eroded in the context of addiction. Oxytocin has also demonstrated the ability to reduce substance use behaviors (e.g., craving, self-administration, tolerance, withdrawal), and improves the neurobiological foundations of AUD. The primary objective of this Stage II study is to test the efficacy of oxytocin versus placebo in improving (1) AUD symptom severity, (2) relationship functioning, and (3) corticolimbic connectivity among couples receiving ABCT therapy.

ELIGIBILITY:
Inclusion criteria

1. Male or female; any race or ethnicity; aged 18-75 years.
2. Able to provide informed consent and function at an intellectual level sufficient to allow accurate completion of the assessment instruments (> 26 on the Mini-Mental State Exam).
3. Married, cohabiting, or in a committed relationship for ≥ 6 months.
4. Identified Patients (IPs) must meet Diagnostic and Statistical Manual of Mental Disorders (DSM-5) diagnostic criteria for current alcohol use disorder. Couples in which both partners meet diagnostic criteria for current Alcohol Use Disorder (AUD) are eligible for participation.
5. Concurrent substance use disorders (e.g., marijuana) are acceptable provided that alcohol is the IP's primary substance of choice.
6. Participants taking psychotropic medications will be required to be maintained on a stable dose for at least four weeks before study initiation. This is because initiation or change of psychotropic medications during the course of the trial may interfere with interpretation of results.

Exclusion criteria

1. Meeting DSM-5 criteria for a history of or current psychotic or bipolar affective disorders, or with current suicidal or homicidal ideation and intent. Those individuals will be referred clinically for treatment.
2. Participants who present a serious suicide risk or are likely to require hospitalization during the study.
3. Participants on psychotropic medications which have been initiated during the past 4 weeks. They may be re-assessed after at least four weeks on a stable dose.
4. Acute alcohol withdrawal as indicated by Clinical Institute Withdrawal Assessment Alcohol Scale Revised (CIWA-Ar) scores >8. They may be re-assessed once they are no longer in withdrawal. Those individuals will be referred for medically supervised detoxification.
5. Severe unilateral intimate partner violence in the past 6 months as defined by the Revised Conflict Tactics Scale (CTS-2).
6. Pregnancy or breastfeeding for women.
7. Individuals with implanted metal devices above the waist will be eligible to enroll in the clinical trial but will not be eligible to participate in the neuroimaging component of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2019-05-16 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julianne Flanagan, PhD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited through internet advertisements, clinician referrals, and flyers. Following preliminary eligibility screening, Identified Patients and partners completed private written informed and a baseline assessment separately for privacy. The baseline assessment included a history and physical (H&P) exam and a battery of standardized self-report and interview measures.
  Recruitment and enrollment occurred from May 2019 to April 2023.
Pre-assignment Details: Participants were 96 adult romantic couples (total N=192) where at least one partner met diagnostic criteria for Alcohol Use Disorder in the past 6 months.Couples were required to have been in their current relationship for at least 6 months. Participants who were taking psychotropic medications were required to be on a stable dose for 4 weeks before enrolling.
Groups:
- Oxytocin: A 40-International Unit (IU) dose of oxytocin self-administered 30 minutes prior to the start of each weekly Alcohol Behavioral Couples Therapy (ABCT) session.
  All participants assigned to 12 weekly, 90-minute therapy sessions delivered by trained Masters or Doctoral-level clinicians consistent with the published manual.
- Placebo: A placebo self-administered 30 minutes prior to the start of each weekly Alcohol Behavioral Couples Therapy (ABCT) session.
  All participants assigned to 12 weekly, 90-minute therapy sessions delivered by trained Masters or Doctoral-level clinicians consistent with the published manual.
Period: Treatment Phase
Arm/Group | Oxytocin | Placebo
Started | 98 | 94
Completed | 78 | 78
Not Completed | 20 | 16
Not completed — Withdrawal by Subject | 9 | 11
Not completed — Lost to Follow-up | 6 | 2
Not completed — Opted out of intervention but completed assessments | 5 | 3
Period: Completed Follow Up Phase (6-month)
Arm/Group | Oxytocin | Placebo
Started | 78 | 78
Completed | 72 | 77
Not Completed | 6 | 1
Not completed — Lost to Follow-up | 6 | 1

BASELINE CHARACTERISTICS:
Groups:
- Oxytocin: A 40-International Unit (IU) dose of oxytocin self-administered 30 minutes prior to the start of each weekly Alcohol Behavioral Couples Therapy (ABCT) session.
  All participants assigned to12 weekly, 90-minute therapy sessions delivered by trained Masters or Doctoral-level clinicians consistent with the published manual.
- Placebo: A placebo self-administered 30 minutes prior to the start of each weekly Alcohol Behavioral Couples Therapy (ABCT) session.
  All participants assigned to 12 weekly, 90-minute therapy therapy sessions delivered by trained Masters or Doctoral-level clinicians consistent with the published manual.
- Total: Total of all reporting groups
Arm/Group | Oxytocin | Placebo | Total
Number analyzed (Participants) | 98 | 94 | 192
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Identified Patient and Partner listed in individual rows.
  years
    Identified Patient: number analyzed (Participants) | 49 | 47 | 96
    Identified Patient | 38.9 (11.8) | 43.3 (12.6) | 41.1 (12.2)
    Partner: number analyzed (Participants) | 49 | 47 | 96
    Partner | 38.6 (13.5) | 42.1 (12) | 40.35 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Identified Patient and Partner listed in individual rows.
  Participants
    Identified Patient: number analyzed (Participants) | 49 | 47 | 96
    Identified Patient: Female | 12 | 14 | 26
    Identified Patient: Male | 37 | 33 | 70
    Partner: number analyzed (Participants) | 49 | 47 | 96
    Partner: Female | 38 | 34 | 72
    Partner: Male | 11 | 13 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 7 | 11
  Not Hispanic or Latino | 94 | 87 | 181
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Identified Patient and Partner listed in individual rows.
  Participants
    Identified Patient: number analyzed (Participants) | 49 | 47 | 96
    Identified Patient: American Indian or Alaska Native | 0 | 1 | 1
    Identified Patient: Asian | 0 | 0 | 0
    Identified Patient: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Identified Patient: Black or African American | 3 | 2 | 5
    Identified Patient: White | 44 | 43 | 87
    Identified Patient: More than one race | 2 | 1 | 3
    Identified Patient: Unknown or Not Reported | 0 | 0 | 0
    Partner: number analyzed (Participants) | 49 | 47 | 96
    Partner: American Indian or Alaska Native | 1 | 0 | 1
    Partner: Asian | 0 | 0 | 0
    Partner: Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
    Partner: Black or African American | 1 | 2 | 3
    Partner: White | 45 | 41 | 86
    Partner: More than one race | 2 | 3 | 5
    Partner: Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Percent Days Abstinent - Measured by Time Line Follow Back (TLFB)
Description: Change in percent days abstinent was measured by the Time Line Follow Back (TLFB), a semi-structured clinical interview that uses calendar prompts to stimulate recall of alcohol consumption. Percent days abstinent (days with no alcohol consumption) were measured at baseline (60 days prior to study entry) and weekly for 12 weeks (end of treatment phase), with lower percentage of drinking days representing better outcomes.
  Time Line Follow Back (TLFB), a clinician assessed measure, will be used to report percent days abstinent (days with no alcohol consumption) and percent days heavy drinking (5 or more days of binge drinking per month).
Time Frame: Baseline to week 12
Measure: Mean (95% Confidence Interval); unit: percentage of days abstinent for alcohol
Groups:
- Oxytocin: A 40-IU dose of oxytocin will be self-administered 30 minutes prior to the start of each weekly ABCT session.
  All participants will receive 12 weekly, 90-minute ABCT therapy sessions delivered by trained Masters or Doctoral-level clinicians consistent with the published manual.
  Oxytocin: A 40-IU dose of oxytocin will be self-administered 30 minutes prior to the start of each weekly ABCT session.
- Placebo: A placebo will be self-administered 30 minutes prior to the start of each weekly ABCT session.
  All participants will receive 12 weekly, 90-minute ABCT therapy sessions delivered by trained Masters or Doctoral-level clinicians consistent with the published manual.
  Placebo: A placebo will be self-administered 30 minutes prior to the start of each weekly ABCT session.
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 49 | 47
percentage of days abstinent for alcohol | 36.8 [25.5 to 48.1] | 35.9 [24.7 to 47.1]

2. Primary Outcome: Change in Relationship Functioning - Measured by Dyadic Adjustment Scale - Short Form (DAS-7)
Description: Change in relationship functioning was measured by the Dyadic Adjustment Scale - Short Form (DAS-7), 7-item Likert-type self-report measure assessing four relationship domains (satisfaction, intimacy, affective expression, and agreement). The DAS-7 was administered at baseline and weekly for 12 weeks (end of treatment). Scores range from 0-36, with higher scores representing better relationship functioning.
Time Frame: Baseline to week 12
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 49 | 47
score on a scale | 25.0 [23.8 to 26.2] | 25.0 [23.7 to 26.2]

3. Primary Outcome: Change in Percent Days Heavy Drinking - Measured by Time Line Follow Back (TLFB)
Description: Change in percent days abstinent was measured by the Time Line Follow Back (TLFB), a semi-structured clinical interview that uses calendar prompts to stimulate recall of alcohol consumption. Percent heavy drinking days defined in a sex-specific manner (> 4 standard drinks for women or > 5 for men) were measured at baseline (60 days prior to study entry) and weekly for 12 weeks (end of treatment phase), with lower percentage of heavy drinking days representing better outcomes.
Time Frame: Baseline to week 12
Measure: Mean (95% Confidence Interval); unit: percentage of heavy drinking days
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 49 | 47
percentage of heavy drinking days | 11.8 [2.3 to 21.2] | 9.9 [0.6 to 19.3]

4. Post Hoc Outcome: Change in Alcohol Problem Severity - Measured by Alcohol Use Disorder Identification Test (AUDIT)
Description: Change in alcohol problem severity was measured by the Alcohol Use Disorder Identification Test (AUDIT), a 10-item Likert-type self-report measure. The AUDIT was administered at baseline and weekly for 12 weeks (end of treatment). Scores range from 0 to 40, with scores of 15 or greater representing moderate to severe Alcohol Use Disorder (AUD).
Time Frame: Baseline to week 12
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 49 | 47
score on a scale | 14.6 [12.9 to 16.4] | 13.1 [11.2 to 14.9]

5. Post Hoc Outcome: Changes in Patient Outcomes Based on Partners' Alcohol Use Disorder (AUD) Status - Measured by Alcohol Use Disorder Identification Test (AUDIT)
Description: Between-group differences in patients' outcomes based on partners' alcohol use disorder (AUD) status measured by the Alcohol Use Disorder Identification Test (AUDIT), a 10-item Likert-type self-report measure. Scores range from 0-40 on the AUDIT, with higher scores representing greater problems with alcohol use, and 15 or greater representing AUD.
  Group differences in patient outcomes included percent days abstinent and percent days heaving drinking, measured by the Time Line Follow Back (TLFB), a semi-structured clinical interview. Outcomes also included patients' relationship functioning, measured by the Dyadic Adjustment Scale-Short Form (DAS-7), a 7-item Likert-type self-report measure, and patients' alcohol problem severity, measured by the AUDIT, a 10-item Likert-type self-report measure.
  DAS score ranges from 0 to 36, with a higher score indicating more positive relationship quality. Scores less than 21 are considered to indicate a relationship in distress.
Time Frame: Baseline to week 12
Measure: Number; unit: Cohen's D
Groups:
- Partner Has Alcohol Use Disorder (AUD): Partners of patients were categorized as having Alcohol Use Disorder (AUD) if they scored 15 or greater on the Alcohol Use Disorder Identification Test (AUDIT)
- Partner Does Not Have Alcohol Use Disorder (AUD): Partners of patients were categorized as not having Alcohol Use Disorder (AUD) if they scored below 15 on the Alcohol Use Disorder Identification Test (AUDIT)
Arm/Group | Partner Has Alcohol Use Disorder (AUD) | Partner Does Not Have Alcohol Use Disorder (AUD)
Number analyzed (Participants) | 48 | 48
Cohen's D
  Percent days abstinent | -0.03 | 0.00
  Percent heavy drinking days | -0.13 | -0.39
  Relationship functioning | -0.04 | 0.01
  Alcohol problem severity | -0.12 | -0.26

ADVERSE EVENTS:
Time Frame: Approximately 9 months (from start of baseline appointment through 12-week treatment phase and 6 month follow up)
Arm/Group | Oxytocin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/98 | 0/94
Serious Adverse Events (participants affected / at risk) | 2/98 | 6/94
Other Adverse Events (participants affected / at risk) | 49/98 | 38/94
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oxytocin (N=98) | Placebo (N=94)
Stroke (Cardiac disorders) | 0 (0) | 1 (1) — with hospitalization
Appendectomy (Surgical and medical procedures) | 0 (0) | 1 (1) — with hospitalization
Hernia surgery (Surgical and medical procedures) | 0 (0) | 1 (1) — with hospitalization
Sepsis (Infections and infestations) | 0 (0) | 1 (1) — with hospitalization
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1) — (pills) with hospitalization
Supraventricular tachycardia/arrhythmia (Cardiac disorders) | 0 (0) | 1 (1) — with hospitalization
Inpatient alcohol detoxification (Psychiatric disorders) | 1 (1) | 0 (0)
Thoracic injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — with hospitalization
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oxytocin (N=98) | Placebo (N=94)
Coronavirus infections (Infections and infestations) | 4 (4) | 11 (11)
Gastrointestinal discomfort (Gastrointestinal disorders) | 16 (22) | 8 (8)
Viral upper respiratory tract infections (Infections and infestations) | 19 (19) | 15 (16)
Headache/Migraine (Nervous system disorders) | 8 (11) | 4 (4)
Injury/Accident (Injury, poisoning and procedural complications) | 10 (11) | 2 (4) — skin burn; burned hand; broken hand; hand wound; finger laceration; facial abrasion; facial contusion; facial scrape; scratched cornea; back injury; torn rotator cuff; broken foot; foot injury; fall resulting in knee/foot abrasions
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 9 (10) | 5 (6)
Influenza (Infections and infestations) | 8 (8) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-03-08): https://cdn.clinicaltrials.gov/large-docs/05/NCT03846505/Prot_SAP_000.pdf
  • Informed Consent Form (2022-08-16): https://cdn.clinicaltrials.gov/large-docs/05/NCT03846505/ICF_001.pdf